CLINICAL TRIAL: NCT01562028
Title: An Open-label Phase II Trial of Erlotinib and Bevacizumab in Patients With Advanced Non-small Cell Lung Cancer and Activating EGFR Mutations
Brief Title: BELIEF (Bevacizumab and ErLotinib In EGFR Mut+ NSCLC)
Acronym: BELIEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 2-11 / MO27911; 2011-004481-15 (EudraCT Number); MO27911 (Other: Roche)
Record Dates: First submitted 2012-03-22; First posted 2012-03-23 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Lung Cancer
Keywords: non small cell lung cancer; advanced; non-squamous; EGFR; mutations
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib plus bevacizumab (Experimental): Patients will be treated with erlotinib and bevacizumab. Bevacizumab: 15 mg/kg i.v. on day 1 of each 3-week cycle (+/- 3 days) Erlotinib: 150 mg p.o., daily
  Interventions: Drug: Erlotinib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Erlotinib — Patients will be treated with erlotinib, 150 mg p.o., daily
  Other Names: Tarceva (R) (Roche)
Drug: Bevacizumab — Patients will be treated with bevacizumab 15 mg/kg i.v. on day 1 of each 3-week cycle (+/- 3 days)
  Other Names: Avastin (R) Roche)

SUMMARY:
Rationale:

Advanced non-small-cell lung cancer (NSCLC) patients harbouring epidermal growth factor receptor (EGFR) mutations (del19 or L858R) show an impressive progression-free survival between 9 and 14 months when treated with erlotinib. However, the presence of EGFR mutations can only imperfectly predict outcome. The investigators hypothesize that progression-free survival could be influenced both by the pretreatment EGFR T790M mutation and by components of DNA repair pathways.

The investigators propose a model of treatment whereby patients with EGFR mutations (single or with T790M) can attain a benefit with longer overall PFS when treated with erlotinib plus bevacizumab. When the patients are grouped by BRCA1 mRNA levels and T790M the hypothesis is that the combination of erlotinib plus bevacizumab can improve the PFS in all subgroups.

DETAILED DESCRIPTION:
Objectives:

1. To determine long-term outcome of patients with advanced non-squamous NSCLC harbouring EGFR mutations with or without T790M mutation at diagnosis and treated with the combination of erlotinib and bevacizumab. Primary endpoint: progression-free survival
2. To evaluate the efficacy and tolerability of the combination
3. To evaluate the correlation of BRCA1 mRNA and AEG-1 mRNA expression and T790M with progression-free survival
4. To monitor EGFR mutations (including T790M) in serum and plasma longitudinally
5. To evaluate molecular biomarkers related to EGFR TKI and bevacizumab

Design:

This is a multinational, multi-center phase II trial of erlotinib plus bevacizumab in patients with advanced non-squamous NSCLC harbouring EGFR mutations confirmed by central re-assessment. Patients will be stratified into two subgroups, with and without EGFR T790M mutation. The stratification will be done after the inclusion of patients.

Sample size: 102 patients

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ECOG performance status 0-2
* Adequate haematological function, coagulation, liver function and renal function
* Pathological diagnosis of predominantly non-squamous, non-small-cell lung cancer (NSCLC)
* TNM version 7 stage IV disease including M1a (malignant effusion) or M1b (distant metastasis), or locally advanced disease not amenable to curative treatment (including patients progressing after radiochemotherapy for stage III disease)
* Measurable or evaluable disease (according to RECIST 1.1 criteria).
* Centrally confirmed EGFR exon 19 deletion (del19) or exon 21 mutation (L858R)

Exclusion Criteria:

* Patients with increased risk of bleeding
* Patients with clinically significant cardiovascular diseases
* Patients with a history of thrombosis or thromboembolism in the 6 months prior to treatment
* Patients with gastrointestinal problems
* Patients with neurologic problems
* Patients who have had in the past 5 years any previous or concomitant malignancy EXCEPT adequately treated basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix or bladder, in situ breast carcinoma.
* Patients with any known significant ophthalmologic anomaly of the ocular surface
* Patients who received prior chemotherapy for metastatic disease
* Patients who received previous treatment for lung cancer with drugs targeting EGFR or VEGF
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2012-06; Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Rosell, MD, Study Chair — Catalan Institute of Oncology, Hospital Germans Trias i Pujol; Stahel Rolf, MD, Study Chair — Laboratory of Molecular Oncology, Clinic of Oncology, University Hospital Zuerich; Miquel Taron, Study Chair — Medical Oncology Service-ICO, Hospital Germans Trias i Pujol
Locations (48):
- France (2):
  - Centre Francois Baclesse, Caen
  - Hôpital de Marseille, Marseille
- Germany (4):
  - Hospital Grosshansdorf, Großhansdorf
  - Thoraxklinik Heidelberg GmbH, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Universitätsklinikum Ulm, Ulm
- Greece (2):
  - University General Hospital of Heraklion, Heraklion
  - Papageorgias Hospital, Thessaloniki
- Ireland (5):
  - St Vincent's University Hospital, Dublin
  - St. James's Hospital, Dublin
  - University Hospital Galway, Galway
  - Mid-Western Regional Hospital, Limerick
  - AMCCH, Tallaght
- Italy (6):
  - Ospedale San Gerardo, Monza
  - Istituto Oncologico Veneto IRCCS, Padua
  - Casa di Cura Maddalena, Palermo
  - Policlinico Tor Vergata Roma, Roma
  - San Camillo Hospital, Roma
  - Policlinico Umberto, Roma
- Spain (11):
  - Hospital General Universitario Alicante, Alicante
  - ICO - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Clínic Barcelona, Barcelona
  - ICO - Girona, Girona
  - ICO - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Clinico Universitario San Carlos, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital General de Valencia, Valencia
  - Hospital La Fe, Valencia
- Switzerland (10):
  - University Hospital Basel, Basel
  - Istituto Oncologica della Svizzera Italiana, Bellinzona
  - Inselspital Bern, Bern
  - Geneva University Hospital, Geneva
  - Fondation du centre Pluridisciplinaire d'Oncologie (CePO), Lausanne
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Onkologiezentrum Berner Oberland, Thun
  - Kantonsspital Winterthur, Winterthur
  - University Hospital Zurich, Zurich
- United Kingdom (8):
  - Mid Essex Hospital Services NHS Trust, Chelmsford, Essex
  - Queen's Hospital, Burton-on-Trent
  - University Hospitals of Leicester, Leicester
  - Royal Marsden Hospital, London
  - Kent Oncology Centre, Maidstone
  - Christie Hospital Manchester, Manchester
  - Wythenshawe Hospital Manchester, Manchester
  - Wrexham Maelor Hospital, Wrexham

REFERENCES:
- [Background] Paez JG, Janne PA, Lee JC, Tracy S, Greulich H, Gabriel S, Herman P, Kaye FJ, Lindeman N, Boggon TJ, Naoki K, Sasaki H, Fujii Y, Eck MJ, Sellers WR, Johnson BE, Meyerson M. EGFR mutations in lung cancer: correlation with clinical response to gefitinib therapy. Science. 2004 Jun 4;304(5676):1497-500. doi: 10.1126/science.1099314. Epub 2004 Apr 29. PMID 15118125
- [Background] Rosell R, Carcereny E, Gervais R, Vergnenegre A, Massuti B, Felip E, Palmero R, Garcia-Gomez R, Pallares C, Sanchez JM, Porta R, Cobo M, Garrido P, Longo F, Moran T, Insa A, De Marinis F, Corre R, Bover I, Illiano A, Dansin E, de Castro J, Milella M, Reguart N, Altavilla G, Jimenez U, Provencio M, Moreno MA, Terrasa J, Munoz-Langa J, Valdivia J, Isla D, Domine M, Molinier O, Mazieres J, Baize N, Garcia-Campelo R, Robinet G, Rodriguez-Abreu D, Lopez-Vivanco G, Gebbia V, Ferrera-Delgado L, Bombaron P, Bernabe R, Bearz A, Artal A, Cortesi E, Rolfo C, Sanchez-Ronco M, Drozdowskyj A, Queralt C, de Aguirre I, Ramirez JL, Sanchez JJ, Molina MA, Taron M, Paz-Ares L; Spanish Lung Cancer Group in collaboration with Groupe Francais de Pneumo-Cancerologie and Associazione Italiana Oncologia Toracica. Erlotinib versus standard chemotherapy as first-line treatment for European patients with advanced EGFR mutation-positive non-small-cell lung cancer (EURTAC): a multicentre, open-label, randomised phase 3 trial. Lancet Oncol. 2012 Mar;13(3):239-46. doi: 10.1016/S1470-2045(11)70393-X. Epub 2012 Jan 26. PMID 22285168
- [Background] Kobayashi S, Boggon TJ, Dayaram T, Janne PA, Kocher O, Meyerson M, Johnson BE, Eck MJ, Tenen DG, Halmos B. EGFR mutation and resistance of non-small-cell lung cancer to gefitinib. N Engl J Med. 2005 Feb 24;352(8):786-92. doi: 10.1056/NEJMoa044238. PMID 15728811
- [Background] Kabbinavar F, Miller VA, Johnson BE, O'Connor P, Soh C-H, ATLAS Investigators. Overall survival in ATLAS, a Phase IIIb trial comparing bevacizumab therapy +/- erlotinib after completion of chemotherapy with bevacizumab for first-line treatment of locally advanced, recurrent, or metastatic non-small cell lung cancer (NSCLC). J Clin Oncol 2010; 28 (May suppl; abstr 7526).
- [Derived] Rosell R, Dafni U, Felip E, Curioni-Fontecedro A, Gautschi O, Peters S, Massuti B, Palmero R, Aix SP, Carcereny E, Fruh M, Pless M, Popat S, Kotsakis A, Cuffe S, Bidoli P, Favaretto A, Froesch P, Reguart N, Puente J, Coate L, Barlesi F, Rauch D, Thomas M, Camps C, Gomez-Codina J, Majem M, Porta R, Shah R, Hanrahan E, Kammler R, Ruepp B, Rabaglio M, Kassapian M, Karachaliou N, Tam R, Shames DS, Molina-Vila MA, Stahel RA; BELIEF collaborative group. Erlotinib and bevacizumab in patients with advanced non-small-cell lung cancer and activating EGFR mutations (BELIEF): an international, multicentre, single-arm, phase 2 trial. Lancet Respir Med. 2017 May;5(5):435-444. doi: 10.1016/S2213-2600(17)30129-7. Epub 2017 Apr 10. PMID 28408243

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 11, 2012 and Oct 28, 2014, 109 eligible patients were enrolled in 29 centers of eight European countries (Spain, Switzerland, UK, Greece, Italy, Ireland, France and Germany). All patients were included in the efficacy analysis.
Groups:
- T790M Positive: Treatment-naive patients with advanced non-small-cell lung cancer positive for an activating EGFR mutation (exon 19 deletion or L858R mutation), with T790M, treated with erlotinib (150 mg p.o., daily) and bevacizumab (15 mg/kg i.v. on day 1 of each 21 day cycle).
- T790M Negative: Treatment-naive patients with advanced non-small-cell lung cancer positive for an activating EGFR mutation (exon 19 deletion or L858R mutation), without T790M, treated with erlotinib (150 mg p.o., daily) and bevacizumab (15 mg/kg i.v. on day 1 of each 21 day cycle).
Period: Overall Study
Arm/Group | T790M Positive | T790M Negative
Started | 37 | 72
Completed | 34 | 70
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T790M Positive | T790M Negative | Total
Number analyzed (Participants) | 37 | 72 | 109
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69.5 [62.3 to 74.0] | 63 [53.4 to 71.2] | 66.1 [57.1 to 72.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 42 | 67
  Male | 12 | 30 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 0 | 7 | 7
  Former smoker | 10 | 20 | 30
  Never smoked | 27 | 45 | 72
Histological diagnosis [Count of Participants; unit: Participants]
  Adenocarcinoma | 34 | 59 | 93
  Adenosquamous carcinoma | 1 | 1 | 2
  Not otherwise specified | 1 | 2 | 3
  Unknown | 1 | 10 | 11
ECOG performance status [Count of Participants; unit: Participants] — ECOG Performance status scaling:
  PS 0:Fully active, able to carry on all pre-disease performance without restriction PS 1:Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work PS 2:Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours PS 3:Capable of only limited self-care, confined to bed or chair more than 50% of waking hours PS 4:Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  Participants
    0 | 17 | 36 | 53
    1 | 18 | 32 | 50
    2 | 2 | 4 | 6
Brain metastasis [Count of Participants; unit: Participants]
  Yes | 7 | 14 | 21
  No | 30 | 58 | 88
Type of EGFR mutation [Count of Participants; unit: Participants]
  Deletion of exon 19 | 23 | 47 | 70
  L858R mutation in exon 21 | 14 | 25 | 39
BRCA1 mRNA expression [Count of Participants; unit: Participants]
  Low (<9.2) | 10 | 13 | 23
  High (≥9.2) | 10 | 13 | 23
  No material or no value | 17 | 46 | 63
AEG1 mRNA expression [Count of Participants; unit: Participants]
  Low (<1) | 11 | 20 | 31
  High (≥1) | 12 | 18 | 30
  No material or no value | 14 | 34 | 48

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Time from the date of enrollment until an investigator-documented progression or death, whichever occurs first.
  Assessment of Progressive Disease (PD) is based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1): at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum recorded on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From the date of enrollment until documented progression or death, whichever occurs first, assessed up to 48 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T790M Positive | T790M Negative
Number analyzed (Participants) | 37 | 72
months | 16 [12.7 to NA] — The upper 95% confidence limit is not estimable, since the number of patients with events is not sufficient. | 10.5 [9.4 to 14.2]

2. Secondary Outcome: Overall Survival
Description: Time from the date of enrollment until death from any cause.
Time Frame: From the date of enrollment until death, assessed up to 48 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T790M Positive | T790M Negative
Number analyzed (Participants) | 37 | 72
months | NA [18.6 to NA] — The median is not reached and the upper 95% confidence limit is not estimable, since the number of patients with events is not sufficient. | 28.2 [21.4 to 41.8]

3. Secondary Outcome: Time to Treatment Failure
Description: Time from the date of enrollment to discontinuation of treatment for any reason including progression of disease (based on RECIST v1.1), treatment toxicity (adverse events classified according to NCI CTCAE version 4.), refusal and death.
Time Frame: From the date of enrollment until discontinuation of treatment, assessed up to 48 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T790M Positive | T790M Negative
Number analyzed (Participants) | 37 | 72
months | 13.4 [5.6 to 19.6] | 8.3 [6.3 to 9.8]

4. Secondary Outcome: Objective Response
Description: Objective response is defined as best overall response (CR or PR) across all assessment time-points during the period from enrollment to termination of trial treatment. Objective response, along with progressive and stable disease, will be determined using RECIST 1.1 criteria:
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters.
  Progression (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum recorded on the trial. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum of diameters recorded on the trial.
Time Frame: Assessed across all time-points from enrollment to termination of trial treatment (max 48 months).
Population: Patients with only 1 tumor assessment are classified as "Non-Evaluable", because they cannot be accounted for the Objective Response rate.
Measure: Count of Participants; unit: Participants
Arm/Group | T790M Positive | T790M Negative
Number analyzed (Participants) | 37 | 72
Participants
  Complete Response | 3 | 3
  Partial Response | 24 | 54
  Stable Disease | 8 | 9
  Progressive Disease | 1 | 3
  Non-Evaluable | 1 | 3

5. Secondary Outcome: Disease Control
Description: Disease control is defined as achieving objective response (CR or PR, across all time-points from enrollment to termination of trial treatment) or stable disease for at least 6 weeks. Objective response, along with SD (disease control) and PD (no disease control), will be determined using RECIST 1.1 criteria:
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters.Progression (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum recorded on the trial. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum of diameters recorded on the trial.
Time Frame: Assessed across all time-points from enrollment to termination of trial treatment (max 48 months).
Measure: Count of Participants; unit: Participants
Arm/Group | T790M Positive | T790M Negative
Number analyzed (Participants) | 37 | 72
Participants
  Disease Control | 35 | 66
  No Disease Control | 2 | 6

6. Secondary Outcome: Duration of Response
Description: Interval from the date of first documentation of objective response (CR or PR) to the date of first documented progression or relapse. Assessment of Objective response and Progressive Disease (PD) is based on the RECIST 1.1 criteria:
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters.
  Progression (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum recorded on the trial. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum of diameters recorded on the trial.
Time Frame: Assessed across all time-points from enrollment to to the date of first documented progression or relapse (max 48 months).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T790M Positive | T790M Negative
Number analyzed (Participants) | 37 | 72
months | NA [14.7 to NA] — The median is not reached and the upper 95% confidence limit is not estimable, since the number of patients with events is not sufficient. | 12 [8.2 to 20.2]

7. Secondary Outcome: Adverse Events
Description: Adverse events graded according to NCI CTCAE V4.
Time Frame: Assessed across all time-points until end of treatment (30 +/-5 days following the last dose of study drug) (max 48 months).
Population: Three patients never started treatment (2 lost to follow-up, one from each arm and 1 withdrawal from T790M negative arm).
Measure: Count of Participants; unit: Participants
Arm/Group | T790M Positive | T790M Negative
Number analyzed (Participants) | 36 | 70
Participants
  Experienced AE/SAE | 36 | 69
  No AE/SAE | 0 | 1
  Experienced SAE | 12 | 19

ADVERSE EVENTS:
Time Frame: Assessed across all time-points until end of treatment (30 +/-5 days following the last dose of study drug) (max 48 months).
Description: One patient from the T790 positive arm never started treatment (lost to follow-up).
  Two patients from the T790 negative arm never started treatment (one lost to follow-up and one withdrawal).
Arm/Group | T790M Positive | T790M Negative
All-Cause Mortality (participants affected / at risk) | 1/36 | 0/70
Serious Adverse Events (participants affected / at risk) | 12/36 | 19/70
Other Adverse Events (participants affected / at risk) | 36/36 | 69/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T790M Positive (N=36) | T790M Negative (N=70)
Thromboembolic event (Vascular disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Appendicitis (Infections and infestations) | 0 | 2
Colonic perforation (Gastrointestinal disorders) | 1 | 1
Confusion (Psychiatric disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2
Lung infection (Infections and infestations) | 0 | 2
Other (Nervous system disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Bone infection (Infections and infestations) | 0 | 1
Bronchial infection (Infections and infestations) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 0 | 1
Other (Gastrointestinal disorders) | 0 | 1
Other (Hepatobiliary disorders) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Other (Musculoskeletal and connective tissue disorders) | 0 | 1
Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Serum amylase increased (Investigations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T790M Positive (N=36) | T790M Negative (N=70)
Hypertension (Vascular disorders) | 33 | 62
Diarrhea (Gastrointestinal disorders) | 30 | 55
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 28 | 55
Proteinuria (Renal and urinary disorders) | 27 | 34
Fatigue (General disorders) | 23 | 34
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 30
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 | 20
Dry skin (Skin and subcutaneous tissue disorders) | 17 | 20
Nausea (Gastrointestinal disorders) | 13 | 20
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 | 18
Mucositis oral (Gastrointestinal disorders) | 15 | 15
Alanine aminotransferase increase (Investigations) | 8 | 21
Anorexia (Metabolism and nutrition disorders) | 10 | 18
Aspartate aminotransferase increase (Investigations) | 7 | 21
Rash acneiform (Skin and subcutaneous tissue disorders) | 10 | 13
Pain (General disorders) | 10 | 12
Other (Skin and subcutaneous tissue disorders) | 9 | 13
Abdominal pain (Gastrointestinal disorders) | 4 | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 13
Headache (Nervous system disorders) | 8 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 15
Constipation (Gastrointestinal disorders) | 8 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 11
Conjunctivitis (Eye disorders) | 9 | 9
Dysgeusia (Nervous system disorders) | 6 | 12
Vomiting (Gastrointestinal disorders) | 7 | 1
Dizziness (Nervous system disorders) | 6 | 10
Paronychia (Infections and infestations) | 8 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 6
Urinary tract infection (Infections and infestations) | 6 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 8
Erythema multiforme (Skin and subcutaneous tissue disorders) | 6 | 6
Other (Eye disorders) | 5 | 7
Upper respiratory infection (Infections and infestations) | 6 | 6
Other (Metabolism and nutrition disorders) | 4 | 7
Other (Gastrointestinal disorders) | 6 | 3
Other (Infections and infestations) | 5 | 5
Depression (Psychiatric disorders) | 2 | 7
Edema limbs (General disorders) | 5 | 4
Fever (General disorders) | 3 | 5
Hemorrhoids (Gastrointestinal disorders) | 4 | 5
Nail infection (Infections and infestations) | 3 | 6
Paresthesia (Nervous system disorders) | 3 | 6
Other (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Anal hemorrhage (Gastrointestinal disorders) | 4 | 3
Dry eye (Eye disorders) | 3 | 5
Dry mouth (Gastrointestinal disorders) | 5 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 6
Oral hemorrhage (Gastrointestinal disorders) | 3 | 5
Thromboembolic event (Vascular disorders) | 2 | 2
Dysphagia (Gastrointestinal disorders) | 4 | 2
Flu like symptoms (General disorders) | 3 | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 5
Other (General disorders) | 3 | 3
Lung infection (Infections and infestations) | 2 | 2
Mucosal infection (Infections and infestations) | 3 | 3
Other (Musculoskeletal and connective tissue disorders) | 1 | 4
Other (Nervous system disorders) | 2 | 2
Anemia (Blood and lymphatic system disorders) | 1 | 4
Anxiety (Psychiatric disorders) | 2 | 3
Bronchial infection (Infections and infestations) | 2 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Creatinine increased (Investigations) | 3 | 2
Hematoma (Vascular disorders) | 2 | 3
Hematuria (Renal and urinary disorders) | 1 | 4
Nail ridging (Skin and subcutaneous tissue disorders) | 2 | 3
Other (Renal and urinary disorders) | 0 | 5
Aphonia (Nervous system disorders) | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Other (Blood and lymphatic system disorders) | 2 | 2
Blood bilirubin increased (Investigations) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Gastritis (Gastrointestinal disorders) | 2 | 2
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 2 | 2
Insomnia (Psychiatric disorders) | 2 | 2
Non-cardiac chest pain (General disorders) | 2 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 3
Rhinitis infective (Infections and infestations) | 1 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 4
Chest pain - cardiac (Cardiac disorders) | 0 | 3
Lip infection (Infections and infestations) | 0 | 3
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 | 1
Oral pain (Gastrointestinal disorders) | 2 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 3
Watering eyes (Eye disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-11-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT01562028/Prot_001.pdf
  • Statistical Analysis Plan (2015-11-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT01562028/SAP_000.pdf